CLINICAL TRIAL: NCT03465189
Title: Validation of a Seizure Monitoring System
Status: Completed | Type: Observational
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: University of Melbourne (Other); Seer Medical (Unknown)
Responsible Party: Principal Investigator, Mark Cook, Principal Investigator, St Vincent's Hospital Melbourne
Other Study IDs: HREC/18/SVHM/50
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Medtronic LINQ Device — Using two LINQ devices that are fixed to scalp to record EEG (in addition to the standard scalp EEG).

SUMMARY:
The investigators aim to determine the feasibility of using the Medtronic LINQ device for epilepsy diagnosis, monitoring and management. The feasibility will be determined by comparing EEG signals from the LINQ system to the gold standard clinical recordings. If seizures can be identified using the LINQ device with the same level of accuracy as adjacent scalp EEG recording electrodes, then the LINQ will be deemed feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epilepsy

Exclusion Criteria:

* Women that are pregnant
* Patients that are highly dependant on medical care
* Patients that cannot give informed consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Verify feasibility of using the LINQ device for epilepsy diagnosis, monitoring and management | one week
  Compare EEG from traditional scalp EEG to the LINQ recordings to determine if seizure activity can be accurately identified

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No